CLINICAL TRIAL: NCT06326567
Title: Comprehensive Connected Cancer Care (C4): Intervention Evaluation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Timothy Mullett (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Timothy Mullett, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MCC-23-MULTI-61; 84032
Record Dates: First submitted 2024-03-15; First posted 2024-03-22 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Cancer; Health Care Utilization
Keywords: Community Programs; Health Equity
MeSH Terms: conditions — Neoplasms; Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Baseline Phase (No Intervention): Each site will complete an 18-month Baseline Phase, in which patients and sites are observed during a period of usual care, prior to introducing the C4 Program intervention. In this phase, a sample of newly diagnosed patients will be recruited and enrolled in the Baseline Group, and data will be collected on them via patient surveys and EHR data abstraction over a period of four months for most outcomes, except for overall survival, which will be assessed at 12 months after diagnosis
- Implementation (Experimental): new sample of newly diagnosed patients (excluding anyone from the Baseline Phase) will be recruited and enrolled in the Implementation Group, and the same data will be collected on them that was collected in the Baseline Group, at the same time points
  Interventions: Other: C4 Program

INTERVENTIONS:
Other: C4 Program — C4 program aims to provide a multi-level intervention program (Patient Level, Healthcare Team and Healthcare System Level) that improves the coordination of care with supportive/ancillary care providers and community services through the use of patient navigation and a digital needs assessment and a closed-loop referral system and improves patient-centered communication and engagement in care through skills training for the healthcare team and provision of culturally appropriate patient educational tools and resources. The program components incorporate three areas that are critical to improving patient-centered care: coordination of care, patient-centered communication and engagement, and psychosocial care and other supportive services.
  Arms: Implementation

SUMMARY:
The C4 program aims to provide a multi-level intervention program (Patient Level, Healthcare Team and Healthcare System Level) that improves the coordination of care with supportive/ancillary care providers and community services through the use of patient navigation and a digital needs assessment and a closed-loop referral system and improves patient-centered communication and engagement in care through skills training for the healthcare team and provision of culturally appropriate patient educational tools and resources. The program components incorporate three areas that are critical to improving patient-centered care: coordination of care, patient-centered communication and engagement, and psychosocial care and other supportive services.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed or recurrent cancer who have not initiated treatment of any kind, including surgery, medical management, and/or radiation
* Patients with one reported social determinants of health (SDOH) need OR patients at high-risk for SDOH needs based on demographic information (racial & ethnic minorities, medicaid/uninsured populations).
* Willingness to provide informed consent to participate

Exclusion Criteria:

* Not able to understand and communicate in English
* Unable and/or unwilling to access the internet on a phone, tablet, or computer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Health Related Quality of Life (FACT-G7) | baseline (enrollment) and 4 months
  The FACT-G7 is a 7-item version of the Functional Assessment of Cancer Therapy-General (FACT-G), a patient-reported outcome measure used to assess health-related quality of life in patients undergoing cancer therapy. The survey assesses the impacts of cancer therapy in four domains: physical, social/family, emotional, and functional. Higher scores represent higher quality of life.

SECONDARY OUTCOMES:
Overall Survival | 12 months
  1 year survival after diagnosis (12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Mullett, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No